CLINICAL TRIAL: NCT05843734
Title: Clinical Performance of Glass Hybrid Restorations in the Treatment of Class III Lesions: A Randomized Clinical Trial
Brief Title: Clinical Performance of Glass-hybrid in the Treatment of Class III Restorations
Acronym: Class-III
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Uzay Koc, Assoc. Prof., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/12-03
Record Dates: First submitted 2022-10-28; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Class III Dental Caries
Keywords: Glass hybrid restorative; Class III; Anterior restoration; FDI criteria

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Equia forte HT (glass-hybrid) group (Experimental): This study planned to investigate the clinical performance of Equia Forte HT (permanent glass hybrid restorative) in the treatment of anterior class III restorations. This arm of the study is the group whose effectiveness was investigated. The results will be evaluated by comparing with a traditional anterior resin composite in terms of functional, biological and aesthetic properties.
  Interventions: Procedure: Equia forte HT
- "G-Aenial anterior" (Active Comparator): This group will serve as a "control". Equia forte HT (glass-hybrid) restorations will compare with the "G-Aenial anterior" anterior resin composite restorations.
  Interventions: Procedure: Equia forte HT

INTERVENTIONS:
Procedure: Equia forte HT — Restoration of anterior class III caries lesions
  Other Names: G-Aenial anterior

SUMMARY:
This is a double blinded, split mouth, randomized clinical study that evaluated the performance of a glass hybrid restorative material in class III lesions. The lesions will be restored with glass hybrid restorative (Equia Forte) or anterior composite resin (G-aenial Anterior). Restorations will be evaluated after 24 months according to FDI criteria and the data will be analyzed.

DETAILED DESCRIPTION:
The aim of this study was to comparatively evaluate the clinical performance of a glass-hybrid-restorative with an anterior composite resin (G-aenial Anterior) in class III lesions.

Participants who are 18 years of age or older and healthy, and who have applied to the Restorative Dentistry Department of Hacettepe University Faculty of Dentistry to receive treatment for class III lesions on their front teeth will be included in the study. After explaining the purpose and conditions of the study, they will be asked to sign an informed consent form. The gender, age, and tooth numbers of the participants to be treated will be recorded. 100 upper incisors of 50 patients will be treated, with attention paid to the balanced distribution of teeth in the right and left arches. The "split-mouth" model will be used in the study, with two teeth included in one mouth and each restorative material placed in one tooth. The restorative material to be placed on the teeth will be determined randomly. Before starting the restoration, papers with the names of both materials will be placed in envelopes, and then the assistant staff will be asked to randomly select one of the envelopes during the restoration stage to provide randomization.Data were will be analyzed with Chi- Square, Fisher's Exact Test, Mann U tests

ELIGIBILITY:
Inclusion Criteria:

* The participant must be at least 18 years of age or older
* The participant has at least two class III lesions and the lesions are in symmetrical teeth located in the right and left arch
* The lesion covers at most 2/3 and at least 1/3 of the dentin
* Participant voluntarily signing the informed consent form
* The participant does not have a physical disability that may prevent them from coming to the control.
* Absence of a periapical pathology in the involved tooth

Exclusion Criteria:

* Having systemic disorders that may prevent the participant from regularly attending treatment and control appointments.
* Having severe periodontal problems in the tooth planned to be treated
* Absence of the opposite of the tooth and not participating in chewing
* Lesions which is limited with the enamel tissue
* Teeth with lesions that are too large to be restored
* Patients with anterior malocclusion
* Patients with parafunctional habits.
* Mentally disabled patients.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Functional properties | 2 years
  The primary factor for determining the clinical performance of a restorative material is the Functional properties. Visual tactile examination tools will be used for evaluating restorations according to FDI criteria by two experienced researchers at 1- week 6-, 12-, 18- and 24- months. The functional properties are scored as 1- clinically excellent, 2-clinically good, 3-clinically sufficient/satisfactory, 4-clinically unsatisfactory 5-clinically poor (replacement necesessry). Clinically 1, 2 and 3 scores are clinical acceptable but 4 and 5 scores are designated as failure.
Esthetic properties | 2 years
  Second outcome is esthetic properties. The secondary factor for determining the clinical performance of a restorative material is the Esthetic properties. Visual examination will be used for evaluating restorations according to FDI criteria by two experienced researchers at 1- week 6-, 12-, 18- and 24- months. The Esthetic properties are scored as 1- clinically excellent, 2-clinically good, 3-clinically sufficient/satisfactory, 4-clinically unsatisfactory 5-clinically poor (replacement necesessry). Clinically 1, 2 and 3 scores are clinical acceptable but 4 and 5 scores are designated as failure.

CONTACTS AND LOCATIONS:
Overall Officials: UZAY Koç VURAL, PhD.DDS, Principal Investigator — Hacettepe
Locations (2):
- Turkey (Türkiye) (2):
  - Hacettepe University School of Dentistry, Ankara
  - Hacettepe University, Ankara

IPD SHARING:
Plan to Share IPD: No